CLINICAL TRIAL: NCT01436110
Title: A Randomised, Double-blind, Double-dummy, Placebo Controlled Multi-centre Study to Evaluate the Efficacy and Safety of Fluticasone Furoate Inhalation Powder and Fluticasone Propionate Inhalation Powder in the Treatment of Asthma in Adults and Adolescents Not Currently Treated With Inhaled Corticosteroids
Brief Title: Clinical Study Evaluating Safety and Efficacy of Fluticasone Furoate and Fluticasone Propionate in People With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115285
Record Dates: First submitted 2011-09-15; First posted 2011-09-19 (Estimated); Results first posted 2014-09-03 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone furoate 50 mcg (Experimental): Once daily inhalation powder via Novel Dry Powder Inhaler
  Interventions: Drug: Fluticasone furoate 50mcg
- Fluticasone propionate 100mcg (Active Comparator): Twice daily inhalation powder via DISKUS/ ACCUHALER
  Interventions: Drug: Fluticasone propionate 100mcg
- Placebo (Placebo Comparator): Inhalation Powder via Novel Dry Powder Inhaler and DISKUS/ ACCUHALER
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone furoate 50mcg — Once daily inhalation powder via Novel Dry Powder Inhaler
  Arms: Fluticasone furoate 50 mcg
Drug: Fluticasone propionate 100mcg — Twice daily inhalation powder via DISKUS/ACCUHALER
  Arms: Fluticasone propionate 100mcg
Drug: Placebo — Inhalation powder via Novel Dry Powder Inhaler and DISKUS?ACCUHALER
  Arms: Placebo

SUMMARY:
A randomised, double-blind, double-dummy, placebo controlled multi-centre study to evaluate the efficacy and safety of fluticasone furoate inhalation powder and fluticasone propionate inhalation powder in the treatment of asthma in adults and adolescents not currently treated with inhaled corticosteroids

DETAILED DESCRIPTION:
This will be a multi-centre, randomised, placebo and active controlled (with rescue medication), double-blind, double-dummy, parallel-group study. Subjects meeting all the inclusion criteria and none of the exclusion criteria during Visit 1 (Screening Visit) will enter a two week Run-in Period. Subjects failing screening will not be eligible for re-screening. During the run-in and double-blind treatment periods subjects will maintain an electronic daily diary to record morning and evening peak expiratory flow (PEF), asthma symptom scores and rescue albuterol/salbutamol use. At Visit 2 (end of run-in/Randomisation Visit), subjects meeting the eligibility criteria will be randomised receive treatment with either fluticasone furoate 50 mcg once daily, fluticasone propionate 100 mcg twice daily or placebo. In addition all subjects will be supplied with albuterol/salbutamol inhalation aerosol to use as required to treat symptoms. Subjects will attend 6 on-treatment visits at Visits 3, 4, 5, 6, 7 and 8 (Weeks 2, 4, 8, 12, 18 and 24 respectively). Subjects will receive treatment for 24 weeks. A follow-up contact will be performed 1-week after completing study medication (Visit 9). Subjects will participate in the study for up to a maximum of 27 weeks (including screening, treatment and follow-up contact).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Outpatient at least 12 years of age with a diagnosis of asthma at least 12 weeks prior to first visit
* Both genders; females of child bearing potential must be willing to use appropriate contraception during the study
* Pre-bronchodilator FEV1 of at least 60% predicted
* FEV1 reversibility of at least 12% and 200ml
* Current asthma therapy that includes a non-corticosteroid controller and/or short acting beta-agonist

Exclusion Criteria:

* History of life-threatening asthma exacerbation with the past 10 years
* Asthma exacerbation requiring oral corticosteroids within the past 3 months or overnight hospital stay within the past 6 months
* Current or recent respiratory infection or current oral candida infection
* Presence of a significant respiratory disease or other medical condition that is uncontrolled or that could affect subject safety or study outcome
* Known or suspected allergy to study medication or materials
* Taking another investigational medication or prohibited medication during the study
* Current smokers or former smokers with significant tobacco exposure
* Previous treatment with fluticasone furoate in a phase II or III study
* Children in Care

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2011-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (20):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Columbia, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brick, New Jersey
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Waco, Texas
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Mexico City
- Netherlands (4):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Hoogwoud
  - GSK Investigational Site, Zutphen
- Peru (3):
  - GSK Investigational Site, Lima, Lima Province
  - GSK Investigational Site, San Miguel, Lima region
  - GSK Investigational Site, Lima
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Wroclaw
- Russia (4):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115285 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants meeting eligibility criteria at the Screening visit entered a 2-week Run-in Period for Baseline safety evaluations and to obtain measures of asthma status. Participants were then randomized to a 24-week Treatment Period. A total of 655 participants were screened; 351 were randomized, and 347 received >=1 dose of study treatment.
Groups:
- Placebo: Participants received placebo via a dry powder inhaler (DPI) once daily (OD) in the evening plus placebo via a different DPI twice daily (BID) for 24 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FF 50 µg OD: Participants received fluticasone furoate (FF) 50 micrograms (µg) inhalation powder via a DPI OD in the evening plus placebo via a different DPI BID for 24 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
- FP 100 µg BID: Participants received fluticasone propionate (FP) 100 µg BID via a DPI plus placebo via a different DPI OD in the evening for 24 weeks. In addition, all participants were provided with albuterol/salbutamol aerosol to be used as rescue medication as needed.
Period: Overall Study
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Started | 116 (These participants were randomized to trial medication.) | 117 (These participants were randomized to trial medication.) | 118 (These participants were randomized to trial medication.)
Intent-to-Treat Population | 115 (These randomized participants received at least a single dose of trial medication.) | 117 (These randomized participants received at least a single dose of trial medication.) | 115 (These randomized participants received at least a single dose of trial medication.)
Completed | 77 | 91 | 95
Not Completed | 39 | 26 | 23
Not completed — Lack of Efficacy | 23 | 14 | 9
Not completed — Withdrawal by Subject | 6 | 8 | 4
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Physician Decision | 3 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Protocol Violation | 3 | 1 | 1
Not completed — Did Not Receive Trial Medication | 1 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID | Total
Number analyzed (Participants) | 115 | 117 | 115 | 347
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.6 (18.03) | 35.4 (14.64) | 36.2 (16.95) | 36.4 (16.57)
Gender [Count of Participants; unit: Participants]
  Female | 81 | 72 | 76 | 229
  Male | 34 | 45 | 39 | 118
Race/Ethnicity, Customized [Number; unit: Participants]
  White - White/Caucasian/European Heritage | 52 | 55 | 54 | 161
  American Indian or Alaska Native | 31 | 30 | 34 | 95
  Mixed Race | 22 | 17 | 18 | 57
  African American/African Heritage | 9 | 14 | 9 | 32
  Asian - East Asian Heritage | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinic Visit Evening (Pre-bronchodilator and Pre-dose) Forced Expiratory Volume in One Second (FEV1) at the End of the 24-week Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Evening clinic visit FEV1 is defined as the clinic visit (pre-bronchodilator and pre-dose) FEV1 measurement taken at the Week 24 clinic visit. Pre-dose and pre-rescue albuterol/salbutamol trough FEV1 were measured electronically by spirometry in the evening at the Baseline through Week 24 clinic visits. The highest of 3 technically acceptable measurements was recorded. Baseline was the pre-dose value obtained at Visit 2. Change from Baseline was calculated as the Week 24 value minus the Baseline value. Analysis was performed using analysis of covariance (ANCOVA) with covariates of Baseline, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing, pre-dose, post-Baseline, on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication. Only those participants with non-missing covariates and post-Baseline FEV1 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 111 | 116 | 112
Liters | 0.089 (0.0331) | 0.126 (0.0323) | 0.191 (0.0328)
Statistical Analysis 1: Comparison: Placebo vs FF 50 µg OD; Test type: Superiority or Other; p = 0.430, ANCOVA; Mean Difference (Final Values) = 0.037, 95% CI 2-sided [-0.055 to 0.128]
Statistical Analysis 2: Comparison: Placebo vs FP 100 µg BID; Test type: Superiority or Other; p = 0.030, ANCOVA; Mean Difference (Final Values) = 0.102, 95% CI 2-sided [0.010 to 0.194]

2. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods Over the 24-week Treatment Period
Description: The number of inhalations of rescue bronchodilator, albuterol/salbutamol inhalation aerosol, used during the day and night was recorded by the participants in a daily electronic diary (eDiary). A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. A 24-hour period was considered as missing if both day time and night time values were missing or if one of the day time or night time values were missing and the other value indicated no use of rescue medication. The Baseline value is the average of the values over the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 114 | 116 | 113
Percentage of rescue-free 24-hr periods | 21.1 (3.20) | 28.9 (3.17) | 31.7 (3.21)

3. Secondary Outcome: Change From Baseline in Daily Evening (PM) Peak Expiratory Flow (PEF) Averaged Over the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the average of the values of the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily trough PM PEF over the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters/minute (L/min)
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 114 | 116 | 113
Liters/minute (L/min) | 7.6 (4.08) | 24.9 (4.04) | 12.0 (4.09)

4. Secondary Outcome: Change From Baseline in Daily Morning (AM) PEF Averaged Over the 24-week Treatment Period
Description: PEF is a measure of lung function and is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each morning and evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 114 | 116 | 113
L/min | 10.8 (3.85) | 30.0 (3.81) | 21.4 (3.86)

5. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods During the 24-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. A 24-hour period was considered as missing if both the day time and night time data were missing or if one was symptom-free but the other was missing. The Baseline value was the average of the values of the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 24-week Treatment Period minus the Baseline value. Analysis was performed using ANCOVA with covariates of Baseline, region, sex, age, and treatment.
Time Frame: From Baseline up to Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 114 | 116 | 113
Percentage of symptom-free 24-hr periods | 16.8 (2.88) | 25.1 (2.85) | 24.3 (2.88)

6. Secondary Outcome: Number of Participants Who Withdrew Due to Lack of Efficacy During the 24-week Treatment Period
Description: The reason for withdrawal was lack of efficacy if a participant was withdrawn due to: clinic FEV1 falling below the FEV1 stability limit; participant experiencing at least 4 days of AM or PM PEF falling below the PEF stability limit and/or at least 3 days of >=12 inhalations/day of albuterol/salbutamol usage during the 7 days immediately preceding any contact; or the occurrence of an asthma exacerbation, defined as the deterioration of asthma requiring the use of systemic (oral, parenteral, or depot) corticosteroids for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. The FEV1 stability limit was calculated as the best pre-salbutamol/albuterol FEV1 at Visit 2 * 80%. The PEF stability limit was calculated as the mean AM PEF from the available 7 consecutive days preceding Visit 2 * 80%.
Time Frame: From the first dose of the study medication until Week 24/Early Withdrawal
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Number analyzed (Participants) | 115 | 117 | 115
Participants | 23 | 14 | 9

ADVERSE EVENTS:
Time Frame: On-treatment adverse events (AEs), defined as those events occurring while participants were on treatment, up to and including the day after the last dose (up to 24 weeks), are reported.
Description: Serious AEs (SAEs) and non-serious AEs were collected in the ITT, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | Placebo | FF 50 µg OD | FP 100 µg BID
Serious Adverse Events (participants affected / at risk) | 3/115 | 0/117 | 1/115
Other Adverse Events (participants affected / at risk) | 36/115 | 38/117 | 39/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | FF 50 µg OD (N=117) | FP 100 µg BID (N=115)
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=115) | FF 50 µg OD (N=117) | FP 100 µg BID (N=115)
Nasopharyngitis (Infections and infestations) | 6 | 8 | 12
Pharyngitis (Infections and infestations) | 10 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 6
Influenza (Infections and infestations) | 4 | 4 | 6
Headache (Nervous system disorders) | 13 | 17 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.